CLINICAL TRIAL: NCT05044338
Title: China Degenerative Valve Disease II Cohort Study (China-DVD2 Study)
Brief Title: Study on Standard Evaluation System and Optimal Treatment Path of Senile Valvular Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yongjian Wu (Other Government)
Responsible Party: Sponsor-Investigator, Yongjian Wu, Chief physician, China National Center for Cardiovascular Diseases
Organization: China National Center for Cardiovascular Diseases (Other Government)
Other Study IDs: 2020YFC2008100
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: imaging — (1) Build the first full information big data cloud platform for diagnosis, treatment and clinical research of senile valvular disease in China (2) To establish a cohort of elderly patients with valvular disease in China and a complete database covering clinical information, functional, imaging evaluation, treatment and follow-up; (3) To analyze the clinical characteristics, functional status and imaging characteristics of senile valvular disease in China, and to understand the current situation of diagnosis and treatment; To establish a whole process standardized comprehensive evaluation system of clinical indicators of senile valvular disease combined with a variety of imaging for Chinese people.

SUMMARY:
The key technology research and standard evaluation system of elderly heart valve disease evaluation is to further establish a domestic multi center and large sample full information big data platform of elderly heart valve disease based on the previous Chinese elderly valve disease cohort and clinical research platform and the national valve disease surgery data platform.

DETAILED DESCRIPTION:
Establish clinical and Imaging Database

ELIGIBILITY:
Inclusion Criteria:

Patients with heart valve disease who are ≥ 65 years old and diagnosed by echocardiography meet the requirements

One of the following criteria:

* (1)Severe mitral stenosis: valve orifice area < 1.0cm2;
* (2)Severe mitral regurgitation: constriction neck width ≥ 7mm, or regurgitation per beat (regurgitation volume)≥ 60ml, or reflux beam area / left atrial area > 50%; Or effective reflux port area (eroa) ≥ 0.4cm2;
* (3)Severe aortic stenosis: mean cross valve pressure difference ≥ 40mmhg, or maximum jet velocity ≥ 4m / s, orValve orifice area < 1.0cm2, it should be differentiated from left ventricular outflow tract stenosis;
* (4)Severe aortic regurgitation: constriction neck width > 6mm, or each pulsation regurgitation ≥ 60ml, or regurgitation Flow fraction ≥ 50%, or jet width ≥ 65% of left ventricular outflow tract, or effective reflux orifice area (eroa) ≥0.3cm2；
* (5)Severe tricuspid stenosis: mean cross valve pressure difference ≥ 5mmhg;
* (6)Severe tricuspid regurgitation: constriction neck width ≥ 7mm, or effective regurgitation orifice area (eroa)≥0.4cm2；
* (7)Severe pulmonary stenosis: the forward blood flow velocity is ≥ 4m / s, which should be differentiated from right ventricular outflow tract stenosis; Severe pulmonary valve regurgitation: massive regurgitation, wide constriction neck

Exclusion Criteria:

* Patients unwilling to accept registration and follow-up;
* Patients with mental illness who cannot cooperate with information collection and follow-up

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Inpatients in each research center
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | Time Frame: 2years
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: yongjian wu, doctor, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mao Y, Liu Y, Zhai M, Jin P, Chen F, Zhang G, Wei L, Liu J, Guo Y, Wu Y, Yang J. Predictors of Paravalvular Leakage After Transcatheter Aortic Valve Replacement in Patients With BAV: A Machine Learning Model. JACC Adv. 2026 Jan 19;5(2):102566. doi: 10.1016/j.jacadv.2025.102566. Online ahead of print. PMID 41558358
- [Derived] Mao Y, Liu Y, Zhai M, Jin P, Li W, Chen F, Yang Y, Zhang G, Liu J, Guo Y, Pan X, Wu Y, Yang J. Clinical significance of machine learning algorithm in predicting PPM during TAVR in small annuli. Cardiovasc Interv Ther. 2026 Jan 5. doi: 10.1007/s12928-025-01215-5. Online ahead of print. PMID 41491442
- [Derived] Mao Y, Liu Y, Zhai M, Jin P, Li W, Dong X, Chen F, Wang X, Wang Y, Zhang G, Li H, Yang Y, Zhang H, Liu J, Guo Y, Wu Y, Xue Y, Zhang J, Frangi A, Yang J. Precision TAVR quantification- AI-accelerated TAVR planning reduces assessment time by 80% in bicuspid aortic stenosis. Eur Heart J Imaging Methods Pract. 2025 Dec 5;3(4):qyaf153. doi: 10.1093/ehjimp/qyaf153. eCollection 2025 Oct. PMID 41445779